CLINICAL TRIAL: NCT00722696
Title: Metabolic Effects of Eccentric Endurance Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vorarlberg Institute for Vascular Investigation and Treatment (Other)
Responsible Party: Heinz Drexel, VIVIT-Institute
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: K01-2008-1
Record Dates: First submitted 2008-07-22; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Metabolism
Keywords: Metabolism; Muscles; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: physical training — 8 weeks of hiking downwards. For the opposite way, a cable car will be used.

SUMMARY:
The purpose of this study is to evaluate metabolic parameters in previously sedentary individuals before and after eccentric endurance training (hiking downwards). Study participants will regularly hike downwards over a difference in altitude of 540 meters during 8 weeks. For the opposite way, a cable car will be used. Metabolic profiles will be obtained at baseline and after the 8 weeks period of eccentric endurance exercise.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age over 18 years

Exclusion Criteria:

* previous systematic endurance training (>3 times per week >30 min)
* body mass index > 35 kg/m²
* heavy smoking (>20 cigarettes per day)
* regular alcohol consumption >60g per day
* history of cardiovascular disease
* established musculoskeletal disease
* unwillingness to stay in the area for the whole period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Change in metabolic parameters during 8 weeks of hiking downwards | 8 weeks

SECONDARY OUTCOMES:
Change in muscle strength during 8 weeks of hiking downwards | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Drexel, Prof, MD., Principal Investigator — Vorarlberg Institute for Vascular Investigation and Treatment (VIVIT-Institute)
Locations (1):
- Vorarlberg Institute of Vascular Investigation and Treatment, Feldkirch, Vorarlberg, Austria